CLINICAL TRIAL: NCT06271655
Title: [BFD-RST-23-004] Rapid Diagnosis of Viral Acute Respiratory Infection to Decrease Unnecessary Antibiotic Utilization in the Emergency Department (RADIATE)
Brief Title: Rapid Diagnosis of Viral Acute Respiratory Infection to Decrease Unnecessary Antibiotic Utilization in the Emergency Department (RADIATE)
Acronym: RADIATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Payette (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor-Investigator, Christopher Payette, Assistant Professor of Emergency Medicine, George Washington University
Organization: George Washington University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BFD-RST-23-004
Record Dates: First submitted 2024-01-05; First posted 2024-02-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Infection; Viral Infection; Upper Respiratory Tract Infections
Keywords: Antibiotic Utilization
MeSH Terms: conditions — Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SPOTFIRE Arm (Experimental): The intervention involves the use of a rapid point-of-care multiplex PCR test to identify viral etiology in patients with acute respiratory illness. This approach aims to provide timely and accurate diagnostic information to guide treatment decisions. Specimen samples will be collected by research staff at the time of ED presentation by NPAAS. Upon collection, the sample will be promptly prepared for testing on the SPOTFIRE R Panel device. In this trial, all providers will view Spotfire results before prescribing antibiotics ; failure to so so will be a protocol violation.
  Interventions: Device: SPOTFIRE R Panel

INTERVENTIONS:
Device: SPOTFIRE R Panel — The intervention involves the use of a rapid point-of-care multiplex PCR test (Spotfire) to identify etiology of patients with ARI. Specimen samples will be collected by research staff at the time of ED presentation. Upon collection, the sample will be promptly prepared for testing on the SPOTFIRE R Panel device. The device will be in the ED to facilitate testing and accelerate delivery of diagnostic results to clinicians. The time when the provider receives the results will be recorded to evaluate the incorporation of results in clinical decision making.

SUMMARY:
The study titled " The Effect of Definitive Identification of Viral Etiology in Emergency Department Patients with Acute Respiratory Infection on Antibiotic Utilization (RADIATE)" aims to investigate the effectiveness of a rapid diagnostic approach in reducing unnecessary antibiotic use in the emergency department (ED) for patients presenting with acute respiratory illness (ARI) due to a virus. Using a prospective design, eligible participants are individuals who visit the ED with complaints related to acute respiratory illness. The study will employ a single-arm consecutive enrollment approach. The intervention involves the implementation of a rapid point-of-care multiplex polymerase chain reaction (PCR) test to promptly identify the viral cause of the infection. By utilizing a rapid diagnostic tool to identify viral etiology, the study aims to provide healthcare professionals in the ED with more accurate information to guide treatment decisions. Ultimately, the goal is to decrease the unnecessary use of antibiotics for ARI's due to a virus, which has several negative outcomes including promotion of antibiotic resistance, exacerbating ED length of stay and encouraging unnecessary additional diagnostic tests.

DETAILED DESCRIPTION:
This prospective single-center, single-arm clinical trial will be conducted to study the initiation of a new diagnostic pathway for acute respiratory illness. After confirming eligibility following ED triage, patients will be enrolled to undergo the Spotfire syndromic assessment (Biomerieux, Inc.). Samples for the test will be collected via a nasopharyngeal swab administered by triage nurse or ED technician in triage. Results from test will be available in approximately 15 minutes. Patients with signs and symptoms of sore throat determined by throat pain or exudates on tonsils will also be tested for Group A streptococcus at enrollment.

Prior to enrollment, the research team asked the initial clinician to delay ordering additional tests until the test was resulted.

Patients who present to the ED with complaints of ARI will be considered eligible for the study. The intervention involves the use of a rapid point-of-care multiplex PCR test (Spotfire) to identify etiology of patients with ARI. Specimen samples will be collected by research staff at the time of ED presentation. Upon collection, the sample will be promptly prepared for testing on the SPOTFIRE R Panel device. The device will be in the ED to facilitate testing and accelerate delivery of diagnostic results to clinicians. The time when the provider receives the results will be recorded to evaluate the incorporation of results in clinical decision making.

For providers who do prescribe antibiotics, the investigators will ask for rationale for antibiotic prescription. Possible causes include: (1) concern for non-respiratory co-infection; (2) concern for respiratory co-infection. (3) patient request; (4) mitigation of legal risk. (5) significant co-morbidities. (6) personal preference / long-standing practice. (7) considered local standard of care. (8) other. In addition to questions above, investigators will specifically ask if physician was more likely to give antibiotics because the viral test was negative.

Patients will also be queried about why they came to the ED including if they had a specific intention to receive antibiotics, additional testing or other reasons.

Both patients and providers will be asked about their confidence in diagnosis, importance of getting results same day.

The investigators will record the time of triage, time of nasopharyngeal swab, time of test results and time communicated with clinician and time that any additional tests are ordered. The results of the test include the presence of any pathogens.

After discharge, patient will receive a chart review, including ICD-10 code, disposition, summary of test results, Strep test ordered and resulted, antibiotics given in ED (and time), ED length of stay, ED discharge, additional diagnostic tests (i.e., chest X-ray, other lab tests.)

The trial was designed to measure the antibiotic prescribing rate for subjects with a definitive viral etiology, a definitive bacterial etiology and no etiology identified. The study team planned an analysis to assess the antibiotic prescribing rate of those with a definitive viral infection versus those with no etiology identified or bacterial origin.

For all consented and tested patients, the investigators will record baseline patient demographics and characteristics. Group data will be compared for equality and inequality of variances, and for non-normality. Continuous variables between groups will be compared by their means using appropriate t-tests after testing for equality of variances. Discrete or categorical variables will be compared between groups by their proportions using chi-square tests. Non-normal data will be tested using non-parametric tests where appropriate. The testing of the difference between groups of some outcome variables will be done with adjustment for their baseline measures. Either an Analysis of Covariance for continuous data or a logistic regression for discrete data will be used as appropriate for these procedures. A minimum significance interval of 0.05 will be used for all comparison tests.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Clinical suspicion of an acute respiratory infection by an emergency department provider
* Patient endorses at least ONE symptom of respiratory illness including: cough, sneezing, runny or stuffy nose, sore throat, headaches, muscle aches, trouble breathing, shortness of breath, fever
* Patient reports symptoms lasting less than 14 days (i.e., no chronic symptoms)
* Patient able to provide informed consent

Exclusion Criteria:

* Patient is a prisoner or ward of state
* Patients that will get antibiotics regardless of of the results of the test (e.g. sepsis, hypoxia, shock, lobar pneumonia, altered mental status, meningitis, pyelonephritis, appendicitis or related, high clinical severity not otherwise specified
* Patients who have tested positive for C. diff in the last 60 days
* Patients who are hospitalized from the emergency department
* Patients that have an oxygen saturation lower than 95% at triage
* Altered mental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Antibiotic Use | Study Enrollment through ED Visit Discharge, up to 24 hours
  The primary outcome measure is the use of antibiotics for treating acute respiratory illness.

SECONDARY OUTCOMES:
Emergency Department Length of Stay | Study Enrollment through ED Visit Discharge, up to 24 hours
  Length of patient stay in the ED from time of arrival to discharge
Utilization of Alternative Tests | Study Enrollment through ED Visit Discharge, up to 24 hours
  Additional diagnostic tests will be measured including chest x-rays, blood laboratory study, urinalysis, antibiotics for non-respiratory infection, anti-viral agents, CT scans
Patient Confidence in Diagnosis | Study Enrollment through ED Visit Discharge, up to 24 hours
  Patient will be asked about their confidence (Not at all confident to Extremely confident) in the diagnosis the day of testing on a Likert scale
Provider Confidence in Diagnosis | Study Enrollment through ED Visit Discharge, up to 24 hours
  Providers will be asked about their confidence in the diagnosis (Not at all confident to Extremely confident) the day of testing on a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Payette, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No